CLINICAL TRIAL: NCT05756725
Title: Improving Cancer Screening and Follow-up in Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Emmons, Professor of Social and Behavioral Sciences, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-1456; R03CA256233-01 (NIH); 3P50CA244433-01S2 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2023-03-06 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Screening; Colorectal Cancer Screening; Implementation
Keywords: Implementation science; Breast cancer screening; Colorectal cancer screening; Abnormal screening followup

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Pilot Sites (Other): All community health centers participating in the study will implement the new population health management tools utilizing tailored implementation strategies
  Interventions: Other: Practice-Level Implementation Strategies

INTERVENTIONS:
Other: Practice-Level Implementation Strategies — The intervention is implementation of new population health management tools that may better leverage patient navigation and other staff resources to ensure timely abnormal follow up of breast and colorectal cancer screening. The research team will work with CHCs to select implementation strategies that will best facilitate integration of the new tools into practice. The team will use electronic health record data (analyzed at the population level) to determine the impact of the new tools on screening outcomes and qualitative data from up to 3 staff and 2 patients per CHC to evaluate integration of the tools into practice.

SUMMARY:
This is an implementation science study that examines implementation of a single intervention and the development of practice-level implementation strategies to facilitate implementation of the intervention.

DETAILED DESCRIPTION:
The research team has a strong partnership with Azara Healthcare, which provides a population management platform to 325 community health centers (CHCs) in 30 US states. This platform, the Data Reporting and Visualization System (DRVS), allows for population- and patient-level tracking and data visualization. Individual CHCs can customize DRVS by using different functionalities that track specific conditions or care gaps. The aim of this study is to pilot test an implementation intervention to integrate new DRVS tools into practice and assess its impact on timely screening and follow-up in health centers based on availability of patient navigators. This is a small, pre-post design pilot test in which the research team will implement screening tools and practice facilitation over a 4-month period and examine rates of screening referrals, screening completion, and diagnostic resolution. The research team will select up to 4 CHCs to participate (two with patient navigation for cancer screening care and two without patient navigation). The CHCs will be selected from among those who use the DRVS system and express interest in the study. As agreed on by sites, the decision to participate in the intervention will be made at the site-level through collaboration with facility leadership and state primary care associations. The intervention is a practice-level clinical strategy that consists of routine care. Participants will be CHC staff whose duties include helping patients to complete cancer screening and follow-up of abnormal tests as well as CHC patients who experience a clinical encounter as a result of use of the tools. As part of the usual DRVS tool roll-out, Azara will provide staff with 1.5 hours of training on use of the new DRVS tools. The research team anticipates using facilitation as an implementation strategy to troubleshoot intervention workflows and to troubleshoot intervention workflows and monitor implementation. However, the team will be evaluating CHC barriers to implementation and may use alternative implementation strategies if warranted. The CHC staff member who interacts with the DRVS in relation to cancer screening will then, as part of the study, participate in 6 hours of facilitation over 4 months to troubleshoot intervention workflows and monitor implementation. The CHC staff who participate in the implementation will be asked to participate in one follow-up, virtual interview. The research team will use coded data to examine the impact of the tools on patient screening outcomes. The team will not have access to the codes that would allow identification (as will be specified in the data use agreement [DUA] with Azara).

The human-subjects research aspect of this project consists of an evaluation of the implementation intervention with up to 3 staff and 2 patients per CHC via one-hour interviews. The CHC staff whose duties include use of the DRVS tools for cancer screening will participate in a semi-structured interview (up to 60 minutes) to assess their experience with the intervention and ideas for further improvements. Patients who interact with the clinic because of the CHCs use of the tools will also participate in a semi-structured interview (up to 60 minutes) to assess their experiences. The CHCs that agree to participate in the study will be informed at the time of their agreement that staff that use the screening tools and patients who have a clinical encounter because of use of the screening tools will be asked to participate in interviews to assess their experience with the tools. Following completion of the pilot intervention test period, the research team will send the designated staff or patient an email invitation to participate in the interview. The email will include a description of the study purpose. Interview questions for staff will cover the use of tools by asking participants to describe how the tools are integrated into their daily practice, as well as perceived barriers and facilitators to using the tools and strategies to overcome barriers. Interview questions for patient participants will cover their experiences with the follow-up and support provided by the CHC staff related to closing their screening gaps. Interviews will be conducted via zoom or the participant's preferred platform. A research assistant will sit in on the interviews to take notes. Interviews will be audio-recorded, and recordings will be saved on a secure HSPH drive. Participants' involvement is complete after the interview.

ELIGIBILITY:
Inclusion Criteria:

* To participate, individuals must be over the age of 18 and employed at a participating Community Health Center.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Number of open orders for FIT screening | 4 months
  Measured from electronic health record
Number of open orders for mammography screening | 4 months
  Measured from electronic health record

SECONDARY OUTCOMES:
Time to diagnostic resolution among those with abnormal FIT tests | 4 months
  Measured from electronic health record
Time to diagnostic resolution among those with abnormal mammograms | 4 months
  Measured from electronic health record
Feasibility of Implementation Strategies | 4 months
  Assessed via Qualitative Interviews
Acceptability of Implementation Strategies | 4 months
  Assessed via Qualitative Interviews
Appropriateness of Implementation Strategies | 4 months
  Assessed via Qualitative Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Emmons, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- United States (3):
  - Coastal Family Health Center, Inc., Biloxi, Mississippi
  - CareSouth Carolina, Inc., Hartsville, South Carolina
  - Partnership Community Health Center, Inc., Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here, after de-identification (text, tables, figures, and appendices). Upon request and appropriate approvals.
Time Frame: Transcripts with no identifiers will be stored on the Harvard Chan shared drive for 7 years. Audio files will be deleted at the end of the study period (expected to be November 2022).
Access Criteria: Outside investigators will need an approved concept proposal to analyze study data and spend the requisite time with study staff to learn about the data elements needed to conduct the proposed analysis. With the assistance from the study's analytic team, s/he will draft a detailed analysis plan and present to the core group of co-investigators. The discussion at this meeting ensures adequate knowledge of the data, and the presenter gains much insight into how the analysis can be most useful and how it relates to previous analyses. Once the plan is approved by this group, it must also be approved by the CHCs that provide the de-identified data. Following approval by the appropriate IRBs and confirmation that it meets HIPAA requirements, s/he may sign a DUA to use a secure, de-identified dataset to complete only the approved analyses and write the manuscript(s) offsite. A formal data analysis plan application and DUA are available. Requests should be directed to jdaly@hsph.harvard.edu.